CLINICAL TRIAL: NCT06581809
Title: Comparative Evaluation of Care Strategies on Dressing Change-induced Bleeding in Patients With Bleeding Malignant Wounds
Brief Title: Comparative Evaluation of Care Strategies on Dressing Change-induced Bleeding in Patients With Bleeding Malignant Wounds (Tumoss)
Acronym: TUMOSS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IC 2023-07
Record Dates: First submitted 2024-08-01; First posted 2024-09-03 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Malignant Wound
Keywords: Malignant wound; Bleeding; Dressing
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: multicenter, open-label/randomized, 2-arm parallel, superiority trial, national.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algosteril (Active Comparator): control arm (Algostéril® hemostatic dressing): dressing used on the day of the bleeding episode in hospital
  Interventions: Other: Algosteril
- Other dressings (Experimental): experimental arm (non-haemostatic dressing): dressing used on the day of the bleeding episode in hospital
  Interventions: Other: Other Dressings: interface, hydrocellular, hydrofiber

INTERVENTIONS:
Other: Algosteril — hemostatic dressing
  Arms: Algosteril
Other: Other Dressings: interface, hydrocellular, hydrofiber — Non-haemostatic dressing
  Arms: Other dressings

SUMMARY:
The goal of this clinical trial is to compare of bleeding on primary dressing removal between a hemostatic dressing and a non-hemostatic dressing positioned following a first bleeding episode. This assessment will be made on adult patient with a malignant wound ≥ 10cm² who presents with a bleeding episode during a hospital consultation.

The primary endpoint is bleeding caused by the removal of a dressing applied during the first bleeding episode observed in the consultation.Effectiveness will be assessed by the resumption of bleeding during the following day's care, in order to respond to 2 care priorities: stopping the bleeding and avoiding its recurrence.The investigators propose a randomized study, with the choice between hemostatic (Algosteril®) or non-hemostatic (interface, hydrocellular, high-absorbency fiber dressing) being randomized and therefore not dependent on the wound or the care team.

In the proposed research, the investigators will evaluate pain on dressing removal, the stress that a bleeding episode can cause, and quality of life in relation to the malignant wound.

The investigators will observe the frequency of bleeding episodes over 6 months, the local care used and the medical management of these bleeding episodes.

In addition, the investigators will pay particular attention to the patient's entourage, as well as to the caregiver who will be carrying out the care, notably by measuring their stress levels during bleeding episodes.

DETAILED DESCRIPTION:
Malignant wounds are the result of the oncogenic process. They may be caused by the initial tumor ulcerating on the skin, or by a secondary localization of the cancer (cutaneous metastasis). They may be external, cavitary or superficial.

The most frequent symptoms are bleeding, odour, pain and exudate. The appearance of these wounds can be impressive for the patient, family and caregivers if they are not used to dealing with this type of wound.

As these wounds are chronic, they need to be managed both in hospital and at home.

A retrospective study carried out at the Institut Curie showed that in 80% of cases, bleeding occurred at the time of treatment.

This bleeding is due to the friable nature of the tissues, which are highly vascularized as a result of tumor angiogenesis. They can therefore bleed easily when the dressing is removed.

The application of an alginate dressing, the only hemostatic dressing reimbursed in towns and cities (in France), seems to increase bleeding on dressing removal, compared with other, non-hemostatic products whose removal is less traumatic (interface, hydrocellular and hydrofiber).

The presence of minor bleeding is not negligible, as it appears to significantly increase the risk of more severe bleeding later on.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and older;
* Carriers of a malignant wound ≥ 10cm²;
* Possibility of participating simultaneously in another research study without an exclusion period at the end of the study;
* Patient having signed an informed consent

Exclusion Criteria:

* Patient under 18 years of age;
* Non-ulcerated nodule, tumor infiltration;
* Patient in the terminal phase of their cancer;
* Patients with a tumor wound that is a cutaneous melanoma;
* Patient refusing to be managed by a private nurse or hospitalization at home (HAD);
* Pregnant or breast-feeding women
* Persons deprived of liberty or under guardianship (including curatorship);
* Persons of legal age under court protection;
* Inability to participate in the study for geographical, social, or psychological reasons.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2025-09-27 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Comparison of bleeding on primary dressing removal between a hemostatic dressing and a non-hemostatic dressing positioned following a first bleeding episode | Day 1 after bleeding
  Bleeding rate on Day 1 of randomization, at the time of dressing change during a first bleeding episode.
  A bleed will be considered as a dressing removal for which the nurse had to:
  * use at least 2 packs of 5 compresses and
  * interrupt her care for > 3 minutes to obtain hemostasis

SECONDARY OUTCOMES:
Assess the pain at D1 when the dressing is removed | Day 1 when the dressing is removed
  Visual Analog Pain Scale (scale from 0 to 10).A higher score indicates greater pain intensity
Observe the frequency of bleeding over 6 months | 6 months
  Number of bleeding episodes over 6 months
Describe the bleeding characteristics and its immediate consequences; | 6 months
  Percent of type of bleeding (sheet or jet / pulsatile bleeding)
Describe local care at the time of a bleeding episode; | 6 months
  Type of the primary dressing used at the time of bleeding (percent)
Assess the stress of patients, family, and caregivers after a bleeding episode | 6 months
  Stress Visual Analogue Scale (scale from 0 (no stress) to 10 (stress maxi))
Wound quality of life | 5 months
  Wound Quality of Life Scale (5 suggested answers per question: not at all, a little, moderately, quite a bit and a lot)
Medical management of bleeding | 6 months
  Description of medical management related to bleeding: treatment initiated or modified; hemoglobin control; Transfusion; hemostatic radiotherapy; surgical or radiological management (embolization); sedation for the refractory symptom of bleeding in end-of-life patients
Assess the bleeding episodes according to the dressing subgroups defined in the nonhemostatic group (Interface and absorbent drainage dressing) | Day 1
  Description of induced bleeding on Day 1 according to the non-hemostatic dressing subgroup

CONTACTS AND LOCATIONS:
Overall Officials: Marguerite NICODEME, Study Director — Institut Curie
Locations (12):
- France (12):
  - EHPAD Laurent Antoine, Agde
  - Hôpital Saint-Loup, Agde
  - Centre François Baclesse, Caen
  - EHPAD Claude Goudet, Marseillan
  - CHU Saint Eloi, Montpellier
  - Groupe Hospitalier Diaconesses Croix Saint Simon, Paris
  - Hôpital Tenon, Paris
  - Institut Curie, Paris
  - CLCC - Institut Godinot, Reims
  - Hôpital Saint Clair, Sète
  - EHPAD Pergolines, Sète
  - EHPAD l'Estagnol, Vias